CLINICAL TRIAL: NCT00241462
Title: Faslodex Observations During Regular Use by Advanced Mammacarcinoma Patients
Acronym: FORUM
Status: Terminated | Type: Observational
Why Stopped: Due to poor patient enrollment
Sponsor: AstraZeneca (Industry)
Other Study IDs: D6997-NL-001; FORUM
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer
Keywords: Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to identify which patients, receiving Faslodex within the approved label, benefit most from Faslodex treatment.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Locally advanced or metastatic hormone sensitive breast cancer with known estrogen receptor (ER) and progesterone receptor (PR) status
* Patient had a recurrence during or after adjuvant anti-oestrogen treatment or progression of the disease during anti-oestrogen treatment

Exclusion Criteria:

* Life threatening metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2005-06; Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Netherlands Medical Director, MD, Study Director — AstraZeneca
Locations (43):
- Netherlands (43):
  - Research Site, Alkmaar
  - Research Site, Almelo
  - Research Site, Almere Stad
  - Research Site, Amsterdam
  - Research Site, Apeldoorn
  - Research Site, Assen
  - Research Site, Bergen op Zoom
  - Research Site, Capelle aan den IJssel
  - Research Site, Delft
  - Research Site, Delfzijl
  - Research Site, Doetinchem
  - Research Site, Dokkum
  - Research Site, Dordrecht
  - Research Site, Drachten
  - Research Site, Ede Gld
  - Research Site, Eindhoven
  - Research Site, Geldrop
  - Research Site, Gorinchem
  - Research Site, Hardenberg
  - Research Site, Heerenveen
  - Research Site, Heerlen
  - Research Site, Hellevoetsluis
  - Research Site, Hilversum
  - Research Site, Hoogeveen
  - Research Site, Leiden
  - Research Site, Leiderdorp
  - Research Site, Leidschendam
  - Research Site, Meppel
  - Research Site, Nieuwegein
  - Research Site, Oss
  - Research Site, Roermond
  - Research Site, Rotterdam
  - Research Site, Stadskanaal
  - Research Site, Terneuzen
  - Research Site, The Hague
  - Research Site, Tilburg
  - Research Site, Utrecht
  - Research Site, Vlaardingen
  - Research Site, Winschoten
  - Research Site, Winterswijk
  - Research Site, Zeist
  - Research Site, Zevenaar
  - Research Site, Zwolle